CLINICAL TRIAL: NCT06448728
Title: Surgical Outcome Studies in Thoracic Wall Reconstruction With Codubix® Ribs
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01132; kt24Appel
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Thoracic
Keywords: Thoracic Wall Reconstruction; Surgical Implantation; Reconstruction Materials; Codubix® Ribs Prosthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to analyze the short- and long-term outcome after surgical implantation of the Codubix® Ribs prosthesis in a descriptive and non-statistical way.

DETAILED DESCRIPTION:
An intact thoracic wall is essential for maintaining organ and respiratory function and upper extremity mobility, and therefore may require surgical intervention if portions of the thoracic wall have been destroyed or removed. Thoracic wall reconstruction is typically needed for cancers originating in or invading the chest wall or for large defects resulting from surgery that removes multiple ribs or the sternum. Less commonly, it is required due to malformations, infections, radiation injuries, or trauma to maintain respiratory function, protect internal organs, and avoid cosmetic defects.

There are several synthetic, metallic, and biologic materials on the market for thoracic wall reconstruction, each with its advantages and disadvantages, and none has proven superior to the others, often being chosen based on the surgeon's experience and preference. Codubix® Ribs, a knitted prosthesis made of polypropylene and polyester yarn, has been used since 2018 for thoracic wall reconstruction due to its high strength, low weight, and non-reactive properties. Moreover, it is radiolucent, easily adjustable to the chest wall's curvature, and maintain enough stiffness to not require additional materials, even for large defects. Although well-established in neurosurgery, its use in thoracic surgery is relatively new and not yet extensively reviewed in literature.

The primary objective is to evaluate the postoperative outcomes after thoracic wall reconstruction with Codubix® Ribs examining mobility, stability, aesthetic outcome and pain. The secondary objectives are to evaluate specific indications for chest wall resection found in the participants and in-hospital complications during the hospital stay.

The results of this study, summarizing our experiences with the relatively unknown prosthesis Codubix Ribs, aim to provide valuable insights and contribute to the broader knowledge base of the medical community regarding effective thoracic wall reconstruction materials.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received full thickness resection of the thoracic wall and reconstruction using Codubix® Ribs
* Patients of all co-morbidities and gender
* Patients that signed written informed consent according to ICH-GCP regulations prior to initiation of any protocol-specific follow-up events
* Patients of age >18 years at the time of informed consent

Exclusion Criteria:

* Patients who have not signed hospital's general consent form for the use of their health-related data for scientific purposes will not be included into the project.
* Patients that received thoracic wall reconstruction with other materials than Codubix® Ribs
* Inability to follow procedures or insufficient knowledge of language
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study collects and evaluates retrospective data of approximately 14 patients who underwent full-thickness thoracic wall resection and reconstruction with Codubix® Ribs starting on February 25th, 2018 up to December 31st, 2023 at the thoracic surgery department of the University Hospital of Basel.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Assessment of mobility | At least 3 months post surgery
  To evaluate mobility of the prosthesis, routine screening for thoracic wall mobility is performed using MRI.
Physical examination | At least 3 months post surgery
  To evaluate the thoracic wall stability and aesthetic outcome, a physical examination is done.
Assessment of disability and symptoms | At least 3 months post surgery
  To assess arm, shoulder and hand disability and symptoms, the QuickDASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire is used. It consists of 11 items that inquire about the individual's ability to perform various activities, such as self-care, work, and recreational activities, as well as the severity of symptoms experienced. It provides a quick and comprehensive assessment of upper extremity function and symptoms, with higher scores on a scale from 0 to 100 indicating greater disability, where 0 represents no disability and 100 represents the most severe disability.
Assessment of pain | At least 3 months post surgery
  To assess the postoperative pain, the Numeric Rating Scale (NRS) is used. The NRS is a commonly used tool for assessing pain intensity,asking the patient to rate their pain on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Details on thoracic wall resection | At least 3 months post surgery
  Information on the thoracic wall resection, including indication, surgical approach and, extend of resection performed are collected.
Risk of mortality | At least 3 months post surgery
  The risk of mortality is evaluated using the Charlson Comorbidity index (CCI). The CCI assigns a score to pre-existing medical conditions, with higher scores on a scale from 0 to 33 indicating a greater burden of comorbidities and a higher risk of mortality.
Number of in-hospital complications | At least 3 months post surgery
  The number of in-hospital complications is assessed using the Clavien-Dindo Classification and CTCAE v5.0 (Common Terminology Criteria for Adverse Events, version 5.0). Both systems grade and classify the severity of adverse events or complications experienced by patients undergoing treatments or surgeries, ranging from ranging from grade I/1 (mild) to grade V/5 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Meret Appel, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinic for Thoracic Surgery, Basel, Canton of Basel-City, Switzerland